CLINICAL TRIAL: NCT02614092
Title: Water-based Activities to Enhance Recall in Veterans (WATER-VET)
Brief Title: Water-based Activity to Enhance Recall in Veterans
Acronym: WATER-VET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1884-P; 12I1-RX001884-01A1 (Other Grant/Funding Number: Department of Veterans Affairs RRD)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; memory impairment; Physical Activity; Exercise; Cognitive Training; Veterans; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Motor Activity | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Water based Activity+ Cognitive Training (Experimental): water-based physical activity + classroom based cognitive training
  Interventions: Behavioral: Water-based Activity + Cognitive Training

INTERVENTIONS:
Behavioral: Water-based Activity + Cognitive Training — This is an 8 month long two phase intervention. The first phase consists of 6 months of thrice weekly pool based physical activity occurring at the Palo Alto VA Health Care System. After completion of the 6 month long water based physical activity, participants transition to a ten session cognitive training program at the Palo Alto VA. The cognitive training classes are approximately two hours in length and will be spread over ten sessions across 4 weeks.

SUMMARY:
This two-year study will evaluate the feasibility of an exercise training augmentation for cognitive training intervention to improve memory performance in Veterans with a diagnosis of amnestic Mild Cognitive Impairment (aMCI). This is a two-phased trial: 1) an exercise phase and 2) a cognitive training program. The exercise phase will be an aquatic based exercise program. A combination of exercise and cognitive training programs designed for persons without cognitive impairment have significantly improved memory more than other single intervention groups (exercise only, cognitive training only) and given the success of combination training programs with healthy older adults, it is important to adapt these programs for persons beginning to exhibit clinically significant memory problems, such as those with aMCI.

DETAILED DESCRIPTION:
The primary research question of the proposed study is this: Is a combination water-based physical exercise + cognitive training program for older Veterans with amnestic Mild Cognitive Impairment (MCI) feasible? The primary aims of the proposed research are: 1) demonstrate adequate recruitment and retention rates; 2) refinement of inclusion/exclusion criteria; and 3) further refine the combination waterbased physical exercise + cognitive training (WATER+CT) intervention.

These aims will be tested in a two-phase clinical trial with a single group design: 1) exercise training phase and 2) a cognitive training phase. The exercise training phase consists of a water-based physical exercise program that emphasizes cardiovascular fitness and strength training through a combination of non-weight bearing exercises that include land-based stretching and water-based activities. This 2-year pilot project will include 50 Veterans diagnosed with amnestic MCI age 50-90. The exercise component consists of a six-month water-based exercise program followed by a four-week cognitive training program. For the first two months of the water-based exercise program, Veterans will come to thrice-weekly group sessions at Aquatic Therapy Center at the VA Palo Alto Health Care System. This will transition to a self-paced exercise program for the remaining four months. After completion of the exercise program, Veterans will begin classroom-based cognitive training at the VA Palo Alto Health Care System (VAPAHCS). The cognitive training is based on an efficacious cognitive program that is structured around two components, pre-training and mnemonic training, both of which have been used successfully in persons with aMCI. Assessments of adherence will be administered throughout treatment and measures of feasibility will be completed post-treatment.

Participants will complete a variety of neuropsychological measures taping into areas of cognition such as attention, executive functioning, and memory. To study possible predictors of treatment response, the investigators will also collect biological (cardiovascular functioning and brain derived neurotrophic factor [BDNF] plasma levels) and genetic data (APOE and BDNF genotypes) from these participants. The investigators hope to provide initial evidence of the feasibility of a waterbased exercise training augmentation for cognitive training thus laying the groundwork for full-scale clinical trials targeting the lessening of cognitive impairment in persons with amnestic MCI by non-pharmacological means.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 50 - 90
* diagnosis of aMCI
* available informant
* at least one musculoskeletal problem
* sufficient visual and auditory acuity to allow neuropsychological testing
* willingness to participate in exercise training +cognitive training program for eight months
* approval of primary provider to participate in an exercise trial

Exclusion Criteria:

* current untreated severe psychiatric disorder, such as:

  * Bipolar I
  * Schizophrenia
  * or Major Depressive Disorder, determined by the Mini International Neuropsychiatric Interview (MINI)
* diagnosis of dementia, Clinical Dementia Rating (CDR) > 0.5; modified Hachinski score 4; or delirium
* history of neurological disorder, e.g.:

  * multiple sclerosis
  * seizure disorder
  * stroke
* history of transient ischemic attacks, or systemic illness affecting central nervous system (CNS) function, e.g.:

  * liver failure
  * kidney failure
  * congestive heart failure
  * systemic cancer
* acute illness or unstable chronic illness e.g., history of severe liver disease

  * cirrhosis
  * esophageal
  * varices
  * ascites
  * portal hypertension
  * hepatic encephalopathy
* current severe cardiac disease, e.g.:

  * uncontrolled atrial fibrillation, defined as mean 24 hour heart rate >85 beats/min, or 24 hour maximal ventricular rate >150 beats/min
  * uncontrolled ventricular arrhythmias, defined as recurrent ventricular tachycardia > 3 beats in succession, or 24 hour packed cell volume (PVC) count > 20%; active
  * pericarditis or myocarditis
  * Class III/IV heart failure and / or ejection fraction < 20%
  * thrombophlebitis
  * pulmonary disease with a drop in O2 Sat with exercise to 90% without oxygen
  * embolism within past six months
* inability to participate in an exercise stress test or inability to exercise consistently because of orthopedic or musculoskeletal problems
* morbid obesity (BMI > 39)
* inability to read, verbalize understanding and voluntarily sign the Informed Consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kaci Fairchild, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After providing informed consent, enrolled participants were screened for eligibility. Only those enrolled participants who met all eligibility criteria were allowed to participate in the water-based activity + cognitive training intervention.
Groups:
- Water Based Activity+ Cognitive Training: This is an 8 month long two phase intervention. The first phase consists of 6 months of thrice weekly pool based physical activity occurring at the Palo Alto VA Health Care System. After completion of the 6 month long water based physical activity, participants transition to a ten session cognitive training program at the Palo Alto VA. The cognitive training classes are approximately two hours in length and will be spread over ten sessions across 4 weeks.
Period: Overall Study
Arm/Group | Water Based Activity+ Cognitive Training
Started | 101
Met All Eligibility Criteria | 31
Completed | 21
Not Completed | 80

BASELINE CHARACTERISTICS:
Arm/Group | Water Based Activity+ Cognitive Training
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 21
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Retention and Recruitment Rates
Description: Feasibility will be demonstrated through ratio of enrolled to completed participants
Time Frame: Through Study Completion, an average of 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Water Based Activity+ Cognitive Training
Number analyzed (Participants) | 31
Participants | 21

2. Secondary Outcome: Change in Delayed Recall of a Word List
Description: Change From Baseline on the Delayed Recall of a Word List at 8 months
Time Frame: Through Study Completion, an average of 8 months
Measure: Mean (Standard Deviation); unit: Words Recalled
Arm/Group | Water Based Activity+ Cognitive Training
Number analyzed (Participants) | 31
Words Recalled | 3.94 (3.94)

3. Secondary Outcome: Participant Adherence to Protocol
Description: Participant completion of study related measurements including pedometers, activity logs, cognitive training homework
Time Frame: Through Study Completion, an average of 8 months
Measure: Mean (Full Range); unit: percentage of weeks completed homework
Arm/Group | Water Based Activity+ Cognitive Training
Number analyzed (Participants) | 31
percentage of weeks completed homework | 63.5 [12.5 to 97.1]

4. Secondary Outcome: Appropriateness of Inclusion and Exclusion Criteria
Description: Number of reported serious and non-serious adverse events reported by participants who were eligible for study participation.
Time Frame: From time of consent until completion of Time 3 assessments, an average of 8 months
Measure: Number; unit: # of events
Arm/Group | Water Based Activity+ Cognitive Training
Number analyzed (Participants) | 31
# of events | 10

ADVERSE EVENTS:
Time Frame: AEs, SAEs, and UAPs were collected from the time of study entry until the end of study participation, an average of 8 months
Description: The definition of AEs and SEs does not differ from the provided definition. AEs and SAEs were collected at each study visit.
Arm/Group | Water Based Activity+ Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 7/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Water Based Activity+ Cognitive Training (N=31)
Cardiac discomfort (Cardiac disorders) | 1 (1) — Chest Tightness that resulted in hospitalization
CVA (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Water Based Activity+ Cognitive Training (N=31)
High Blood Pressure (Cardiac disorders) | 3 (5)
Low Blood Pressure (Cardiac disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The final participant completed cognitive training in a remote environment due to COVID19 shelter-in-place orders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02614092/Prot_SAP_000.pdf